CLINICAL TRIAL: NCT05904834
Title: Effect of a Flexibility Program on the Extensibility of the Hamstrings and the Thoracic and Lumbar Spinal Curvatures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Esparza Ros, Director of the International Kinanthropometry Chair, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20092013
Record Dates: First submitted 2023-05-22; First posted 2023-06-15 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Spine Injury; Hamstring Injury; Lumbar Hyperlordosis; Kyphosis
Keywords: Flexibility training; Dancers; Ballet; Flexibility testing
MeSH Terms: conditions — Spinal Injuries; Swayback; Kyphosis

STUDY DESIGN:
Intervention Model Description: Single intervention group and single control group
Who Masked: Investigator
Masking Description: The investigators on charge of the test do not know the group they are measuring
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flexibility training (Experimental): The intervention group will undergo a flexibility training focused on hamstring extensibility. Each will they will take part in four stretching sessions besides the normal dance training.
  Interventions: Other: Flexibility training
- No training (No Intervention): The control group will continue with their training routine during the experiment.

INTERVENTIONS:
Other: Flexibility training — Each session consisted of three or four exercises, of which three were static stretches and if there was a fourth, it was dynamic. The duration of each exercise was 20 seconds with 15 seconds rest between sets and 30 seconds rest between exercises.
  Arms: Flexibility training

SUMMARY:
The goal of this clinical trial is to analyse the effect of an intervention program based on hamstring flexibility on the extensibility and curvatures of the spine in dancers.

Participants will be dance student with ten years of experience that will undergo a program of stretching four times per week during seven weeks, followed by a detraining period, and a retraining period of three weeks. There will be a pre-test, a post-test and two re-tests after the intervention.

The results will be compared with a control group of dancers that will not take part in the stretching program.

DETAILED DESCRIPTION:
Four measurements were carried out, one before the intervention (pre-test), one after the first stretching programme (post-test), one after a short period of detraining (re-test 1) and the last one at the end of a second period of intervention (re-test 2), analysing the intra-group and inter-group differences for each of the dependent variables.

The sample components (n=61) were divided into two groups following a random distribution carried out by an external researcher. The intervention group (IG), which consisted of 31 dancers, underwent the hamstring stretching programme for a first period of 7 weeks and a second period of 3 weeks after a short period of detraining. The intervention consisted of static and dynamic stretching of the hamstring muscles 4 days per week. The control group (CG), composed of 30 dancers, did not perform the stretching programme. Both groups attended their practical classes in the conservatory. During the detraining period the dancers of both groups took a break from physical exercise.

The variables measured are hamstring extensibility and sagittal spine disposition and pelvic tilt.

ELIGIBILITY:
The inclusion criteria were:

1. students enrolled for at least 18 ECTS credits at the High Conservatory of Dance;
2. previous experience of 10 years in dance;
3. practice dance at least 4 days a week;

(c) not suffer from any chronic pathology or at the time of the study; (d) not practising any other physical exercise apart from dance.

Exclusion criteria:

1. Not attending at least 80% of the practical sessions of the Conservatory throughout the programme;
2. being pregnant at the beginning of the study or getting pregnant during the development of the study;
3. having undergone surgery on the spine or hamstring musculature;
4. having suffered a hamstring injuries in the last year or during the study;
5. having structured spinal disorders;
6. having an injury at the time of the assessment that prevents her from taking the measurements;
7. stretching of the hamstring musculature outside the conservatory.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Linear hamstring flexibility | Pre-test (week 1)
  The flexibility of the hamstring will be assessed with different linear test. Sit and reach test will be performed and the measure will be reported in centimeters
Linear hamstring flexibility | Post-test (week 8)
  The flexibility of the hamstring will be assessed with different linear test. Sit and reach test will be performed and the measure will be reported in centimeters
Linear hamstring flexibility | Re-test 1 (week 11)
  The flexibility of the hamstring will be assessed with different linear test. Sit and reach test will be performed and the measure will be reported in centimeters
Linear hamstring flexibility | Re-test 2 (week 14)
  The flexibility of the hamstring will be assessed with different linear test. Sit and reach test will be performed and the measure will be reported in centimeters
Angular hamstring flexibility | Pre-test (week 1)
  The flexibility of the hamstring will be assessed with angular tests. Straight leg raise will be performed in the active and passive versions and the result will be reported in grades
Angular hamstring flexibility | Post-test (week 8)
  The flexibility of the hamstring will be assessed with angular tests. Straight leg raise will be performed in the active and passive versions and the result will be reported in grades
Angular hamstring flexibility | Re-test 1 (week 11)
  The flexibility of the hamstring will be assessed with angular tests. Straight leg raise will be performed in the active and passive versions and the result will be reported in grades
Angular hamstring flexibility | Re-test 2 (week 14)
  The flexibility of the hamstring will be assessed with angular tests. Straight leg raise will be performed in the active and passive versions and the result will be reported in grades
Thoracic spinal curvatures | Pre-test (week 1)
  The thoracic spinal curvatures will be assessed in different positions, including relaxed standing, the sit and reach test and Macrae & Wright test. The result will be reported in grades.
Thoracic spinal curvatures | Post-test (week 8)
  The thoracic spinal curvatures will be assessed in different positions, including relaxed standing, the sit and reach test and Macrae & Wright test. The result will be reported in grades.
Thoracic spinal curvatures | Re-test 1 (week 11)
  The thoracic spinal curvatures will be assessed in different positions, including relaxed standing, the sit and reach test and Macrae & Wright test. The result will be reported in grades.
Thoracic spinal curvatures | Re-test 2 (month 14)
  The thoracic spinal curvatures will be assessed in different positions, including relaxed standing, the sit and reach test and Macrae & Wright test. The result will be reported in grades.
Lumbar thoracic spinal curvatures | Pre-test (week 1)
  The lumbar spinal curvatures will be assessed in different positions, including relaxed standing, the sit and reach test and Macrae & Wright test. The result will be reported in grades.
Lumbar thoracic spinal curvatures | Post-test (Week 8)
  The lumbar spinal curvatures will be assessed in different positions, including relaxed standing, the sit and reach test and Macrae & Wright test. The result will be reported in grades.
Lumbar thoracic spinal curvatures | Re-test 1 (week 11)
  The lumbar spinal curvatures will be assessed in different positions, including relaxed standing, the sit and reach test and Macrae & Wright test. The result will be reported in grades.
Lumbar thoracic spinal curvatures | Re-test 2 (Week 14)
  The lumbar spinal curvatures will be assessed in different positions, including relaxed standing, the sit and reach test and Macrae & Wright test. The result will be reported in grades.
Pelvic Tilt | Pre-test (week 1)
  The pelvic tilt will be assessed in different positions, including relaxed standing, the sit and reach test and Macrae & Wright test. The result will be reported in grades.
Pelvic Tilt | Post-test (Week 8)
  The pelvic tilt will be assessed in different positions, including relaxed standing, the sit and reach test and Macrae & Wright test. The result will be reported in grades.
Pelvic Tilt | Re-test 1 (week 11)
  The pelvic tilt will be assessed in different positions, including relaxed standing, the sit and reach test and Macrae & Wright test. The result will be reported in grades.
Pelvic Tilt | Re-test 2 (Week 14)
  The pelvic tilt will be assessed in different positions, including relaxed standing, the sit and reach test and Macrae & Wright test. The result will be reported in grades.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No
Personal information is not going to be shared under any circumstances. Only unidentified and impersonal information will be used.